CLINICAL TRIAL: NCT03130348
Title: Phase II Study of Ibrutinib With or Without Bortezomib and Dexamethasone for the Treatment of Patients With Relapsed/Refractory Immunoglobulin Light Chain Amyloidosis
Brief Title: Ibrutinib With or Without Bortezomib and Dexamethasone in Treating Patients With Relapsed or Refractory Immunoglobulin Light Chain Amyloidosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was dropped at site before participation
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1687; NCI-2017-00660 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1687 (Other: Mayo Clinic in Florida); P30CA015083 (NIH)
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Amyloidosis; Immunoglobulin Light Chain Deposition
MeSH Terms: conditions — Amyloidosis | interventions — Bortezomib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ibrutinib, bortezomib, dexamethasone) (Experimental): Patients receive ibrutinib PO QD on days 1-28. After 3 courses, patients who achieve partial response repeat treatment every 28 days for up to 18 courses in the absence of disease progression or unacceptable toxicity. Patients who do not achieve partial response after 3 courses continue receiving ibrutinib PO QD on days 1-28. Beginning at course 4, patients who do not achieve partial response also receive bortezomib SC and dexamethasone PO on days 1, 8, and 15. Treatment repeats every 28 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Ibrutinib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well ibrutinib with or without bortezomib and dexamethasone works in treating patients with immunoglobulin light chain amyloidosis that has come back after a period of improvement or that does not respond to treatment. Ibrutinib and bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ibrutinib with or without bortezomib and dexamethasone may work better in treating patients with relapsed or refractory immunoglobulin light chain amyloidosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the overall hematologic response rate (stringent complete response [sCR] + amyloid complete response [ACR]+ very good partial response [VGPR] + partial response [PR]) during the first 6 cycles for ibrutinib with bortezomib and dexamethasone added for lack of response in patients with amyloid light chain (AL).

SECONDARY OBJECTIVES:

I. To evaluate overall hematologic response rate (sCR+ACR+VGPR+PR) of single agent ibrutinib in patients with AL.

II. To evaluate overall hematologic response rate (sCR+ACR+VGPR+PR) to ibrutinib + bortezomib and dexamethasone (Vd) in subjects with progressive disease after initial response to single agent ibrutinib.

III. To describe the toxicities associated with ibrutinib, alone and in combination with Vd, in patients with AL.

IV. To determine the organ response in AL patients treated with ibrutinib alone and in combination with Vd.

V. To determine 3 year progression free survival of AL patients on the study.

TERTIARY OBJECTIVES:

I. To characterize health related quality of life of patients. II. To determine the caregiver and patient disease burden. III. To determine the correlation between cardiac biomarkers and hematologic response to therapy.

IV. To evaluate the effect of ibrutinib on AL microenvironment. V. To characterize BTK expression in neoplastic plasma cells. VI. To evaluate the characterization of CD38 expression on neoplastic plasma cells.

OUTLINE:

Patients receive ibrutinib orally (PO) daily (QD) on days 1-28. After 3 courses, patients who achieve partial response repeat treatment every 28 days for up to 18 courses in the absence of disease progression or unacceptable toxicity. Patients who do not achieve partial response after 3 courses continue receiving ibrutinib PO QD on days 1-28. Beginning at course 4, patients who do not achieve partial response also receive bortezomib subcutaneously (SC) and dexamethasone PO on days 1, 8, and 15. Treatment repeats every 28 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, and then every 6 months for 2 years.

ELIGIBILITY:
Criteria:

* Measurable disease of AL amyloidosis as defined by at least ONE of the following:

  * Serum monoclonal protein >= 1.0 by protein electrophoresis
  * > 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Free light chains (abnormal absolute value, ratio and the dFLC > 5 mg/dL)

Inclusion Criteria:

* Histological diagnosis of AL amyloidosis as based on detection by polarizing microscopy of green birefringent material in Congo red-stained tissue specimens; the type must have been confirmed unequivocally
* Must have had one prior line of systemic therapy for AL; Note: patients who do not achieve at least a PR to frontline therapy in 3 months may be eligible after discussion with study chair
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 100,000/mm^3 or >= 50,000/mm^3 if bone marrow involvement independent of transfusion support in either situation
* Hemoglobin >= 8.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) unless due to Gilbert's syndrome or of non-hepatic origin
* Aspartate transaminase (AST) =< 3 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) =< 3 x ULN
* Creatinine =< 3 mg/dL and creatinine clearance (CrCL) >= 25 ml/min
* Negative serum pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only
* Ability to complete questionnaire(s) by themselves or with assistance
* Ability to provide written informed consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Willing to provide bone marrow and blood samples for correlative research purposes

Exclusion Criteria:

* Any of the following:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception; Note: persons of childbearing potential and persons able to father a child who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials; subjects must agree to not donate sperm during and after the study; for persons of childbearing potential, these restrictions apply for 1 month after the last dose of study drug; for persons able to father a child, these restrictions apply for 3 months after the last dose of study drug
* Concomitant high dose corticosteroids (concurrent use of corticosteroids) while on single agent ibrutinib; EXCEPTION: patients may be on chronic steroids (maximum dose 20 mg/day prednisone equivalent) if they are being given for disorders other than amyloid, (i.e., adrenal insufficiency, rheumatoid arthritis, etc)
* Active malignancy =< 3 years prior to registration; EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix; Note: if there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Known history of human immunodeficiency virus (HIV) or active hepatitis C virus or active hepatitis B virus infection or any uncontrolled active systemic infection
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk
* Receiving any other investigational agent which would be considered as a treatment for AL amyloidosis
* Vaccinated with live, attenuated vaccines =< 4 weeks prior to registration
* Clinically overt multiple myeloma (i.e. original hypercalcemia, renal failure, anemia, bone lesions [CRAB] criteria); Note: extent of marrow plasmacytosis is not prohibitive
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction =< 6 months prior to registration, or any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* NT-ProBNP > 8,500 pg/mL
* Use of strong and moderate CYP3A inhibitors and inducers =< 7 days prior to registration
* Anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon); Note: use of low molecular weight heparin (or any anticoagulation agent) is allowed provided there is no history of bleeding (minor or major) =< 12 months prior to registration; the treating physician should discuss the case with the study chair
* History of stroke or intracranial hemorrhage =< 6 months prior to registration
* Known central nervous system metastasis
* Major surgery or a wound that has not fully healed =< 4 weeks prior to registration
* Surgery or invasive procedure requiring sutures or staples for closure =< 7 days prior to registration
* Minor procedures (such as a central line placement, needle biopsy, thoracentesis, or paracentesis) =< 3 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-15 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Overall hematologic response rate during the first 6 courses for patients treated with ibrutinib, bortezomib, and dexamethasone | Up to 6 months
  Will include a confirmed stringent complete response, amyloid complete response, very good partial response, and partial response. Confirmation will be defined as a response that is maintained on two consecutive evaluations at least 2 weeks apart. Progression will be defined as either hematologic or organ progression. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 3 years
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. Adverse events will be summarized separately for single agent Ibrutinib and combination therapy.
Organ response rate | Up to 3 years
  Will be estimated by the total number of patients who have an organ response divided by the total number of evaluable patients who had involvement in that organ at baseline. Exact binomial 95% confidence intervals for the true organ Up to response rate will be calculated.
Overall hematologic response rate for single agent ibrutinib | Up to 6 months
  Will be estimated by the total number of patients who achieve a partial response, very good partial response, stringent complete response, or amyloid complete response while receiving single agent ibrutinib divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true overall hematologic response rate will be calculated.
Progression-free survival | From registration to the earliest date of documentation of disease progression (on single agent or combination therapy) or death due to any cause, assessed up to 3 years
  Will be estimated using the method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Taimur Sher, Principal Investigator — Mayo Clinic